CLINICAL TRIAL: NCT02005835
Title: Improving Uptake and Retention in PMTCT Services Through Novel Approaches in Family Supported Care and in Community Peer Outreach Support in Malawi
Brief Title: Promoting Uptake and Retention of Option B+ in Malawi
Acronym: PURE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lighthouse Trust (Other)
Collaborators: World Health Organization (Other); AIDS Fonds (Other); Mothers2Mothers (Unknown); Kamuzu University of Health Sciences (Other); Management Sciences for Health (Other); Dignitas International (Other); University of North Carolina, Chapel Hill (Other); University of Malawi (Other); Ministry of Health and Population, Malawi (Other Government)
Responsible Party: Principal Investigator, Sam Phiri, PhD, MSc, DCM, Executive Director, Lighthouse Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PUREMalawi
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: HIV
Keywords: HIV; Option B+; Prevention of Mother to Child Transmission

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Facility-based Peer Support (Other): Facility-based Peer Support to provide the following at the clinic
  * Routine standard clinical care based on the MoH guidelines
  * Mentor mothers provide education and psychosocial support at facility
  * Weekly support groups provided in clinic
  * Phone call, SMS, or home visit for each missed appointment
  Interventions: Other: Facility-based Peer Support
- Community-based Peer Support (Other): Community-based Support from Peer Mothers (Expert mothers):
  * Routine standard clinical care based on the MoH guidelines
  * Mentor mothers provide education and psychosocial support in community prior to each visit
  * Monthly support groups in community
  * Home visits for each missed appointment
  Interventions: Other: Community based peer support
- Standard of Care (No Intervention): The Standard of care as outlined in the Malawi HIV integrated Care Guidelines

INTERVENTIONS:
Other: Community based peer support — Community-based Support from Peer Mothers (Expert mothers):
  Routine standard clinical care based on the MoH guidelines Mentor mothers provide education and psychosocial support in community prior to each visit Monthly support groups in community Home visits for each missed appointment
  Arms: Community-based Peer Support
Other: Facility-based Peer Support — Facility-based Peer Support to provide the following at the clinic
  Routine standard clinical care based on the MoH guidelines Mentor mothers provide education and psychosocial support at facility Weekly support groups provided in clinic Phone call, SMS, or home visit for each missed appointment
  Arms: Facility-based Peer Support

SUMMARY:
The purpose of this study is to determine if enhanced support for women and their families within facilities and/or through community outreach will result in improved retention in the continuum of PMTCT care.

DETAILED DESCRIPTION:
The Malawi Ministry of Health (MoH) has embarked on a novel and ambitious programme to prevent mother to child transmission of HIV (PMTCT) known as "Option B Plus". This programme takes a public health approach to promote maternal health and eliminate paediatric HIV infections through a "test and treat" model, offering all HIV-infected pregnant and breastfeeding women lifelong ART regardless of CD4 count or clinical stage. The overall goal is to improve ART uptake and retention, and thus outcomes, of HIV-infected pregnant women and their infants in the continuum of ART services.

Although the Option B Plus strategy offers an attractive rapid ART scale-up alternative to the WHO PMTCT recommendations and has the potential to profoundly impact maternal and infant outcomes, it has not been implemented in any programme setting. Operational challenges throughout the cascade of PMTCT services may affect the uptake and adherence to highly active ART treatment (HAART) by pregnant women, the follow-up of HIV-exposed infants and the long-term retention of this patient population. Several issues identified at the national level are potential threats to the successful implementation and scale up of Option B plus: a) potential suboptimal uptake of HAART by asymptomatic pregnant women due to low treatment literacy and stigma; b) low adherence to HAART and poor follow-up of HIV exposed infants; and c) lack of psycho-social support for long term retention in this relatively asymptomatic patient population (Schouten et al. 2011).

The aim of the overall project (4 years) is to evaluate facility-based and community-based support models to strengthen uptake and retention of mothers and families in PMTCT care in Malawi. Our hypothesis is that enhanced support for women and their families within facilities and/or through community outreach will result in improved retention in the continuum of PMTCT care.

We will conduct a cluster randomized clinical trial evaluating three support models for the implementation of the Option B+ program. Each of the 21 clinics will be randomized to one of the three adherence and support strategies. Arm 1 is the standard of care arm as outlined by the Ministry of Health, Arm 2 is facility level support by a peer educator and Arm 3 is community level support by a peer educator.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected women Presenting for Antenatal Care, Labor&Delivery, or post-partum Infants of Enrolled mothers Husbands/Spouses of Enrolled mothers

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Retention in Care | 12 months post ART initiation
  The primary outcome is the proportion of women retained alive and on ART at 12 months post ART initiation.

SECONDARY OUTCOMES:
Retention at 24 months | 24 months post ART initiation
  The proportion of Women alive and retained on ART at 24 months post ART initiation
Child HIV status | 6 weeks, 12 months, 24 months
  Children tested at 6 weeks, 12 months, and 24 months
HIV free survival | 6 weeks, 12 months, 24 months
  HIV-free infant survival at 6-weeks, 12 months and 24 months
Family retention | 12 months
  Partner/family involvement, including: a) husband/children tested for HIV; b. eligible husbands/children who start ART; c. husband/children engaged in care at 12 months
Maternal Viral Load | 6 months and 2 years post ART initiation
  Proportion of women with HIVRNA <1000 copies at 6 months and 2 years post initiation
Maternal resistance | 6 months, 2 years
  Of women failing ART, the proportion with HIV drug resistance
Infant HIV resistance | 6 weeks, 12 months, 24 months
  Of HIV infected infants, the proportion with HIV drug resistance
Social outcomes | 12, 24 months
  Social outcomes, including impact of task shifting on burden of care in facilities, quality of life for patients and their families, disclosure and shifts in boundaries of professional and lay care for lay health care workers as assessed by mixed methodology.

OTHER OUTCOMES:
Economics | baseline, 12, 24 months
  Economic indicators including cost effectiveness ratios of support models, equity of access to PMTCT services by geographic area, socio-economic profiles of mothers and families accessing care to assess equity, and indicators for health system impacts such as time at work, overtime, number and types of cases treated, motivation and satisfaction by health workers as assessed by mixed methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Phiri, PhD, MSc., Principal Investigator — Lighthouse Trust
Locations (1):
- Ministry of Health Facilities, Lilongwe, Malawi

REFERENCES:
- [Derived] van Lettow M, Tweya H, Rosenberg NE, Trapence C, Kayoyo V, Kasende F, Kaunda B, Hosseinipour MC, Eliya M, Cataldo F, Gugsa S, Phiri S; PURE Malawi consortium. Baseline characteristics of study sites and women enrolled in a three-arm cluster randomized controlled trial: PMTCT uptake and retention (pure) Malawi. Reprod Health. 2017 Jul 11;14(1):82. doi: 10.1186/s12978-017-0343-0. PMID 28693525
- [Derived] Cataldo F, Sam-Agudu NA, Phiri S, Shumba B, Cornelius LJ, Foster G. The Roles of Expert Mothers Engaged in Prevention of Mother-to-Child Transmission (PMTCT) Programs: A Commentary on the INSPIRE Studies in Malawi, Nigeria, and Zimbabwe. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S224-S232. doi: 10.1097/QAI.0000000000001375. PMID 28498193
- [Derived] Hosseinipour M, Nelson JAE, Trapence C, Rutstein SE, Kasende F, Kayoyo V, Kaunda-Khangamwa B, Compliment K, Stanley C, Cataldo F, van Lettow M, Rosenberg NE, Tweya H, Gugsa S, Sampathkumar V, Schouten E, Eliya M, Chimbwandira F, Chiwaula L, Kapito-Tembo A, Phiri S; PURE Malawi Consortium. Viral Suppression and HIV Drug Resistance at 6 Months Among Women in Malawi's Option B+ Program: Results From the PURE Malawi Study. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2(Suppl 2):S149-S155. doi: 10.1097/QAI.0000000000001368. PMID 28498184
- [Derived] Phiri S, Tweya H, van Lettow M, Rosenberg NE, Trapence C, Kapito-Tembo A, Kaunda-Khangamwa B, Kasende F, Kayoyo V, Cataldo F, Stanley C, Gugsa S, Sampathkumar V, Schouten E, Chiwaula L, Eliya M, Chimbwandira F, Hosseinipour MC; PURE Malawi Consortium. Impact of Facility- and Community-Based Peer Support Models on Maternal Uptake and Retention in Malawi's Option B+ HIV Prevention of Mother-to-Child Transmission Program: A 3-Arm Cluster Randomized Controlled Trial (PURE Malawi). J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S140-S148. doi: 10.1097/QAI.0000000000001357. PMID 28498183
- [Derived] Cataldo F, Chiwaula L, Nkhata M, van Lettow M, Kasende F, Rosenberg NE, Tweya H, Sampathkumar V, Hosseinipour M, Schouten E, Kapito-Tembo A, Eliya M, Chimbwandira F, Phiri S; PURE Malawi Consortium. Exploring the Experiences of Women and Health Care Workers in the Context of PMTCT Option B Plus in Malawi. J Acquir Immune Defic Syndr. 2017 Apr 15;74(5):517-522. doi: 10.1097/QAI.0000000000001273. PMID 28045712
- [Derived] Chiwaula LS, Chirwa GC, Cataldo F, Kapito-Tembo A, Hosseinipour MC, van Lettow M, Tweya H, Kayoyo V, Khangamwa-Kaunda B, Kasende F, Trapence C, Gugsa S, Rosenberg NE, Eliya M, Phiri S; PURE Malawi Consortium. The value of informal care in the context of option B+ in Malawi: a contingent valuation approach. BMC Health Serv Res. 2016 Apr 19;16:136. doi: 10.1186/s12913-016-1381-y. PMID 27095249